CLINICAL TRIAL: NCT06458660
Title: LinkPositively+ An Enhanced Mobile Health App Delivered Intervention to Improve HIV Care Outcomes Among Black Women Affected by Mental Health and Violence
Brief Title: LinkPositively+ A Mobile Health App Delivered Intervention to Improve HIV Care Outcomes Among Black Women Affected by Mental Health and Violence
Acronym: LPP Plus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guiding Right, Inc. (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IN-US-985-7186
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: HIV/AIDS; Mental Health Issue
Keywords: HIV, AIDS, Mindfulness Meditation, Women, Care Continuum, mobile app, Violence,
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm: LinkPositively (Active Comparator): Women assigned to the LinkPositively arm will have access to all four components of the LinkPositively app. Women will be scheduled for a session with staff to inform them of their assigned virtual Peer Navigator (PN). Staff will train participants on how to download the app, explain the five components, using each component, and contacting their PN. Within the first week after, virtual PNs will complete a one-on-one, in-person or phone intake session with the participant, based on the participant's preference. During this intake session, the PN will conduct a participant needs assessment to connect her to HIV medical care via local health clinics and identify other areas of need, services of need, and assisted referrals (domestic violence services, mental health care, substance abuse treatment, housing and legal support, etc.). PNs will provide trauma-informed emotional and informational support, including guidance on accessing information about referred services.
  Interventions: Behavioral: LP
- Intervention Arm: LinkPositively+ (Experimental): Women assigned to the LPP+ arm will receive all components of the LP arm plus access to mindfulness videos via the app, in addition to participating in a virtual 6-session weekly, PN led mindfulness meditation enhanced intervention. The sessions will be delivered in real time, by PNs and will involve 1 on 1 discussions on a) the principles and health benefits of mindfulness meditation, b) lived experiences of women living with HIV and intersectional identities of being Black, and doubling identifying as women, c) experiencing trauma in personal relationships, d) ethnic pride, e) sex/gender pride, and f) positive self-affirmations. Sessions will be conducted online, in-app, and include culturally congruent video clips, role playing, and skills building activities that enhance self-pride and coping during stressful situations.
  Interventions: Behavioral: LPP+: Mindfulness Meditation Delivered

INTERVENTIONS:
Behavioral: LPP+: Mindfulness Meditation Delivered — During the 6-week intervention period, participants will receive reminder SMS text messages at a time selected by the participant at 48 and 24-hrs before each scheduled study visit. Within 24 hours after every session, participants will receive an SMS text reminder to complete a session satisfaction survey. If the satisfaction surveys are not completed within 48 hours after each session, participants will receive an additional SMS text message once per day for three consecutive days after each planned study visit. Twenty-four hours before each scheduled study visit after study visit number 1, participants will an SMS text requiring a one-character response (1= yes, 2=no), asking if participants practiced any mindfulness meditation techniques since the last session. Participants who have not interacted with the app during the previous week will receive an accountability call to assess barriers to participation.
  Arms: Intervention Arm: LinkPositively+
Behavioral: LP — LinkPositively is a culturally tailored, trauma-informed smartphone app for Black women living with HIV/AIDS affected by interpersonal violence. Core components of LinkPositively include: a) Virtual Peer Navigation that includes phone and text check-ins and 4 weekly one-on-one video sessions to build skills to cope with barriers and navigate care; b) Social Networking platform to receive peer support; c) Educational and Self-care database with healthy living and self-care tips; d) GPS-enabled Resource Locator for HIV care and ancillary support service agencies; and e) ART self-monitoring and reminder system.
  Arms: Control Arm: LinkPositively

SUMMARY:
The investigative team will conduct a 2-arm randomized control trial to examine the preliminary effect of LinkPositively+ (LPP) an enhanced version of LinkPositively (LP) mobile app on improved HIV care outcomes including improved retention in HIV care, ART adherence, and viral suppression using hair sample analysis and passive electronic, medical record review, and secondarily, self-reported increased social support via activation of social support networks (i.e., assessed by utilization), self-efficacy, and utilization of ancillary support services at baseline, 3- and 6-month post enrollment. Black women living with HIV (WLHA) with a lifetime history of interpersonal violence, who have been linked to care but may have fallen out of care in the past year will be randomized 1:1 to either the LP arm or the LPP arm.

DETAILED DESCRIPTION:
In the US, Black WLHA are less likely to be engaged in care and adherent to antiretroviral therapy (ART) than other racial groups. Black women account for 61% of diagnoses among all women; only 56% are retained in care and 49% are virally suppressed. HIV disparities are also observed in Oklahoma state, where Black women have HIV diagnosis rates that are 8 times higher than White women. Interpersonal violence; defined as physical, sexual, and/or psychological abuse by a male intimate or non-intimate partner disproportionately affects Black women and is associated with poor outcomes along the HIV care continuum. The confluence of co-occurring adverse mental health and socio-structural barriers (e.g., HIV stigma, medical mistrust) further contribute to poor HIV care outcomes. Social support through informal peer networks and Peer Navigators have been successful in improving HIV care among WLHA, by increasing self-efficacy and offsetting socio-structural barriers. NIMH-funded LinkPositively (LP) is a pilot-tested, culturally-tailored, trauma-informed mHealth intervention responsive to interpersonal violence for Black women. LP aims to improve HIV care outcomes including improved retention in HIV care, ART adherence, and to ultimately achieve viral suppression among Black WLHA residing in EHE jurisdictions (California and Oklahoma) from baseline and 3- and 6-month post enrollment visits. It is hypothesized that this is achieved through increased social support and activation of social support networks, self-efficacy, and utilization of ancillary support services. App components include a social networking platform, education and self-care tips, resource locator, and ART self-monitoring and reminders. Participants of LP have expressed unaddressed mental health symptoms indicative of depression and/or PTSD. Mindfulness meditation has demonstrated success as a stress management tool to mitigate negative mental health outcomes. Given this, we plan to add and test a mental health component within the LP app for Black WLHA (known as LinkPositively+) to support Black WLHA in addressing mental health symptoms indicative of depression and/or PTSD that negatively affect sustained engagement in HIV related care and treatment.

ELIGIBILITY:
Inclusion Criteria: a) aged 18 years or older, b) cisgender or transgender woman, c) as Black or African American racial/ethnic identity, d) Living with HIV/AIDS, e) able to read, speak, and understand English, e) ever-experienced physical, sexual, and/or psychological abuse by a current or former partner of non-partner, and f) owner of a smartphone with internet browsing capabilities.

-

Exclusion Criteria: a) Unwillingness to participate in the study, b) cognitive impairment that would limit participation with study procedures, c) Male Gender, d) HIV negative serostats

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as a woman
Enrollment: 60 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Preliminary effect of LPP+ to improve HIV care outcomes | 3- and 6-month Post Baseline
  The study aims to examine the preliminary effect of LPP+; mindfulness meditation plus PN plus LP app (e.g., social networking platform, education and self-care tips, resource locator, and ART self-monitoring and reminders) to improve HIV care outcomes including improved retention in HIV care, ART adherence, and viral suppression using empirical hair sample analysis (ART adherence) and passive electronic health medical review (viral suppression).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Guiding Right, Inc., Oklahoma City, Oklahoma
  - New Hope Wellness Center, Oklahoma City, Oklahoma
  - Guiding Right, Inc., Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No
No current plan.